CLINICAL TRIAL: NCT05659277
Title: The Physiological, Psychological, and Cognitive Effects of Workplace Stress, SelfManagement Habits, and Irregular Shift Hours on First Responders
Brief Title: The Effects of Stress & Irregular Shift Hours on First Responders
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Endominance (Industry)
Collaborators: Dr. John J. Ratey (Unknown); F1RST Clinic (Dr. Heather Twedell) (Unknown); HEM Pharma Inc. (Industry); iMediSync (Unknown)
Responsible Party: Sponsor
Other Study IDs: 10433
Record Dates: First submitted 2022-11-07; First posted 2022-12-21 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Workplace Stress; Mental Health; HRV; EEG; PTSD
Keywords: First Responder; Shift Work; PHQ9; GAD7
MeSH Terms: conditions — Occupational Stress; Psychological Well-Being; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples will be lab processed and analyzed for the diversity of gut bacteria, dietary habits as well as gut microbiota-derived metabolites from exogenous dietary substrates and endogenous host compounds. Individual results will not be provided.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Workplace Stress and Irregular shift hours — The physiological, psychological, and cognitive impacts that workplace stress and irregular shift hours have on first responders.

SUMMARY:
First Responders are expected to maintain high-performance levels under extreme conditions. However, constant intense workplace stress, physical work demands, and irregular shift hours are taking a severe toll on frontline workers. These demands often lead to physical and mental health problems, poor job performance, and lifestyle issues. Without better support and resources, these demands will continue to cause first responders to be trapped in a vicious cycle that typically includes occupational trauma, stress, and maladaptive coping skills.

The purpose of this research is to:

1. Better understand the physiological, psychological, and cognitive impacts workplace stress and irregular shift hours have on first responders
2. Better understand the most prominent challenges first responders face when trying to manage their own physical and mental health.

Through the results of this study, we hope to identify possible solutions/interventions at the individual, clinical and departmental levels to help first responders better manage their stress and improve their quality of life.

DETAILED DESCRIPTION:
This study aims to expand and improve current research regarding the physiological, psychological, and cognitive impacts that workplace stress and irregular shift hours have on first responders. The investigators will examine electroencephalogram (EEG)/heart rate variability (HRV) measurements and gut microbiota to help bridge the connection between the impacts of a physically and mentally demanding workplace with highly irregular shift hours on first responders. There are numerous studies conducted to evaluate how stress impacts first responders in areas such as physical and mental health, but there lacks comprehensive research that examines the physiological, psychological, and cognitive impacts of workplace stress and irregular shift hours have on first responders in the U.S.

There also lacks information of the challenges first responders face when trying to manage their physical and mental health. To conduct these objectives, we will focus on these specific aspects:

1. The impact of shift hours (especially longer shift hours, e.g., firefighters 24 vs. 48 shift hours) on first responders, specifically in connection to sleep disorders and other cognitive function-related issues.
2. The connection between workplace incidents and stress/alertness levels - even during off-duty hours.
3. First responder self-help/stress relief coping techniques or modalities and their efficacy

ELIGIBILITY:
Inclusion Criteria:

* Full-Time, actively employed First Responder
* Participants must be 18 years of age and older
* Participants must be able to read and write English
* Participants must be able to provide consent independently
* Participants must provide a legitimate postal address/P.O Box
* Participants must have access to a device such as a computer or a smartphone

Exclusion Criteria:

* Unable to provide a stool sample due to health status or functional impairment
* Unable to complete EEG measurement due to health status
* Cognitively impaired persons
* Department volunteers
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First Responders including firefighters, police, SWAT, EMTs, detectives, and dispatchers.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-04-11 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
aMCI (Amnestic Mild Cognitive Impairment) via Electroencephalogram (EEG) | up to 3 months
  Using an advanced wireless EEG device, PPG is measured using the following frequency bands for the prediction of aMCI: Absolute power of delta(1-4Hz), alpha1(8-10Hz), beta2(15-20Hz), beta3(20-30Hz), gamma(30-45Hz) and relative power-delta (1-4Hz), theta (4-8Hz), alpha1 (8-10Hz), alpha2 (10-12Hz), beta1 (10-15Hz), beta2(15-20Hz) and gamma(30-45Hz).
  Specially trained machine learning algorithms can process quantitative EEG to identify subtle evidence of aMCI, thus enabling early interventions that have the greatest potential for delaying or preventing the progression of aMCI to Alzheimer's disease.
  Individual results will be provided.
Brain Functionality via Electroencephalogram (EEG) | up to 3 months
  PPG is measured using the following frequency bands for the prediction of brain functionality: Absolute power of delta(1-4Hz), alpha1(8-10Hz), beta2(15-20Hz), beta3(20-30Hz), gamma(30-45Hz) and relative power-delta (1-4Hz), theta (4-8Hz), alpha1 (8-10Hz), alpha2 (10-12Hz), beta1 (10-15Hz), beta2(15-20Hz) and gamma(30-45Hz).
  3D brainwave analysis highlights the functional, rather than the structural, status of key brain areas, offering special insights into cortical dysfunction or compensatory activity. This brain map highlights areas where the balance between slow (theta, 4-8Hz) waves and fast (beta, 15-20Hz) waves differs from that expected based on age and sex-matched normal healthy population. Lower-than-expected levels of function are reported along with higher- than expected levels.
  Individual results will be provided.
ANS (Autonomic Nervous System) stress analysis via simultaneous Electroencephalogram (EEG) and HRV (heart rate variability) | up to 3 months
  The stress report analyzes ones PPG rhythm pattern with an AI algorithm, displaying 5 stages of stress from homeostasis to burnout (homeostasis, alarm, resistance, exhaustion, and burnout). HRV indicates balance between the activity of the two branches of the ANS.
  Individual results will be provided.

SECONDARY OUTCOMES:
Cognitive Orientation & Social-Emotional Competency Assessment (COSEC) | up to 3 months
  An online cognitive propensity and behavioral preference diagnostic tool. COSEC is designed to understand people's various tendencies that occur during the process between perceiving the environment and responding in action. It illustrates an individual's personality and aptitude as an outcome shaped by their environment and the perception of the world around them. COSEC incorporates the environmental impact on the individual by looking at the unique process of a person's perception, conception, and behavior process. Assessments are scored using an algorithm to generate quantified measurements based on multifactorial relationships between a subject's responses.
  Participants who complete the study will receive their personalized digital report called the COBI report.

OTHER OUTCOMES:
Microbiome Analysis | up to 3 months
  Investigators will analyze participants' microbiomes to better understand diet habits and lifestyles. Enrolled participants will receive an at-home stool sample kit with instructions for the collection, storage, and shipping of samples. Samples will be lab processed and analyzed for the diversity of gut bacteria, dietary habits as well as gut microbiota-derived metabolites from exogenous dietary substrates and endogenous host compounds. Individual results will not be provided.
Health and Lifestyle survey | up to 3 months
  Demographic, health, and lifestyle data.
Depression Scores - Patient Health Questionnaire (PHQ-9) | up to 3 months
  PHQ-9 is a self-administered, 9-question diagnostic tool that rates depression using 9 DSM-V criteria for depression based on mood. Each of the 9 DSM-V criteria is scored as "0" (not at all) to "3" (nearly every day). Higher scores indicate greater severity of depressive symptoms. Individual results will not be provided.
Anxiety Scores - Generalized Anxiety Disorder (GAD-7) | up to 3 months
  GAD-7 is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. The GAD-7 items include 1) nervousness; 2) inability to stop worrying; 3) excessive worry; 4) restlessness; 5) difficulty in relaxing; 6) easy irritation and 7 fear of something awful happening. Higher scores indicate greater severity of anxiety symptoms. Individual results will not be provided.
Post-traumatic stress syndrome (PTSD) - PCL-5 | up to 3 months
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of post-traumatic stress syndrome (PTSD). Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4: "0" (not at all) to "4" (extremely). A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 score between 31-33 is indicative of probable PTSD. Individual results will not be provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Endominance Inc., Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research Study Landing Page — https://www.endominance.com/fr2.0